CLINICAL TRIAL: NCT01212341
Title: A Phase I Study of Allogeneic NK Cell Therapy in Patients With Refractory/Relapsed Lymphoma or Solid Tumor
Brief Title: Allogeneic Natural Killer (NK) Cell Therapy in Patients With Lymphoma or Solid Tumor
Acronym: MG4101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: GC Biopharma Corp (Industry)
Responsible Party: Tae Min Kim/Assistant Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MG4101_P1
Record Dates: First submitted 2010-09-18; First posted 2010-09-30 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Malignant Lymphomas; Solid Tumors
Keywords: Allogenetic NK cells; Lymphomas; Solid tumors
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Singe-dose infusion (Experimental): Cohort 1: 1x10^6 cells/kg Cohort 2: 1x10^7 cells/kg
  Interventions: Biological: Allogeneic NK cells
- Repeated dose infusion (Experimental): Cohort 3: 1x10^6 cells/kg Cohort 4: 3x10^6 cells/kg Cohort 5: 1x10^7 cells/kg Cohort 6: 3x10^7 cells/kg
  Interventions: Biological: Allogeneic NK cells

INTERVENTIONS:
Biological: Allogeneic NK cells

SUMMARY:
Allogeneic natural killer (NK) cells (MG4101) were manufactured from normal healthy donor who underwent leukapheresis. These cells were processed based on a novel method for ex vivo activation and expansion using an irradiated and activated autologous feeder cell system. MG4101 has anti-tumor activities against various tumors including malignant lymphomas in vitro as well as in vivo tumor model.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Histologically or cytologically confirmed malignant lymphoma or solid tumor
* After the failure of standard treatment
* KPS >70 or ECOG PS 0-2
* Adequate bone marrow, renal, and liver functions
* Expected survival at least 3 months
* Informed consent

Exclusion Criteria:

* Pregnancy or lactating woman
* HIV patients
* Prior exposure to cell-based therapy
* Hypersensitivity to interleukin-2
* Patients with autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To determine the MTD of allogenetic NK cells | 4-5 weeks
  DLT is defined as follows:
  * Any toxicity at grade 3 or over for 5 days or more
  * All grade 4 toxicities
  * GVHD at grade 2 or over

SECONDARY OUTCOMES:
To determine the overall response rate | 4-5 weeks
  RECIST v1.1 for solid tumor or revised response criteria for malignant lymphoma
To evaluate the safety | 4 -5 weeks
  NCI-CTCAE v3.0
To evaluate the pharmacokinetics of allogeneic NK cells | 4-5 weeks
  To quantify the persistence of donor NK cells in recipients

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea